CLINICAL TRIAL: NCT02984787
Title: 3D Versus 2D Laparoscopic Total Gastrectomy With Spleen-preserving Splenic Hilum Lymph Nodes Dissection for Advanced Proximal Gastric Cancer: A Randomized Controlled Trial
Brief Title: 3D Versus 2D Laparoscopic Total Gastrectomy With Splenic Hilum Lymph Nodes Dissection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Deputy Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Experiment20161201
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Splenic Hilum Lymph Nodes Dissection
Keywords: Gastric Cancer; 3D; 2D
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D Laparoscopic total gastrectomy (Experimental): Participants including in the 3D laparoscopic total gastrectomy (3D-LTG) group will undergo 3D-LTG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: 3D Laparoscopic total gastrectomy
- 2D Laparoscopic total gastrectomy (Active Comparator): Participants including in the 2D laparoscopic total gastrectomy (2D-LTG) group will undergo 2D-LTG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: 2D Laparoscopic total gastrectomy

INTERVENTIONS:
Procedure: 3D Laparoscopic total gastrectomy — When participants with advanced proximal gastric cancer are randomized in the 3D laparoscopic-assisted totalgastrectomy (3D-LTG) group, they will received 3D-LTG with spleen-preserving splenic hilum lymph nodes dissection
  Other Names: 3D-LTG
  Arms: 3D Laparoscopic total gastrectomy
Procedure: 2D Laparoscopic total gastrectomy — When participants with advanced proximal gastric cancer are randomized in the 2D laparoscopic-assisted totalgastrectomy (2D-LTG) group, they will received 2D-LTG with spleen-preserving splenic hilum lymph nodes dissection
  Other Names: 2D-LTG
  Arms: 2D Laparoscopic total gastrectomy

SUMMARY:
The investigators will perform a prospective randomized comparison between 3D and 2D laparoscopic total gastrectomy with splenic hilum lymph nodes dissection.

DETAILED DESCRIPTION:
A prospective randomized comparison of 3D and 2D laparoscopic surgery for advanced gastric cancer with spleen-preserving splenic hilum lymph nodes dissection will be performed, to evaluate the safety and feasibility for the extensive application of the novel 3D laparoscopic technique. The evaluation parameters are number of group No.10 lymph nodes harvested, perioperative clinical efficacy, postoperative life quality and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

1. Primary proximal gastric adenocarcinoma confirmed pathologically by endoscopic biopsy;
2. cT2-4aN0-3M0 at preoperative evaluation according to AJCC Cancer Staging Manual, 7th Edition.
3. Eastern Cooperative Oncology Group (ECOG): 0 or 1;
4. American Society of Anesthesiologists （ASA） score: Ⅰto Ⅲ;
5. Written informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Severe mental disorder;
3. Previous upper abdominal surgery (except laparoscopic cholecystectomy);
4. Previous gastrectomy, endoscopic mucosal resection, or endoscopic submucosal dissection;
5. Enlarged or bulky regional lymph node diameter larger than 3 cm based on preoperative imaging;
6. Other malignant disease within the past 5 years;
7. Previous neoadjuvant chemotherapy or radiotherapy;
8. Contraindication to general anesthesia (severe cardiac and/or pulmonary disease);
9. Emergency surgery due to a complication (bleeding, obstruction, or perforation) caused by gastric cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of splenic hilum lymph nodes harvested | 7 days

SECONDARY OUTCOMES:
Early complication rate | 30 days
  The early complication rate is defined as the event observed during operation and within 30 days after surgery.
Operative time | Intraoperative
  It will be assessed with the unit of "minute".
Operative blood loss | Intraoperative
  It will be assessed with the unit of "ml".
Time of splenic hilum lymph nodes dissection | Intraoperative
  It will be assessed with the unit of "minute"
Number of total lymph nodes harvested | 7 days
Poster-operative recovery course | 30 days
  Time to first ambulation (unit of hour), flatus (unit of hour), liquid diet (unit of hour) and duration of hospital stay (unit of day) are used to assess the postoperative recovery course.
Quality of life | 1 year
  It will be assessed with questionnaire of "WHO-QOL-100" (WHO was short for world health organization)
3-year disease free survival rate | 3 years
3-year overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, Principal Investigator — the Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No